CLINICAL TRIAL: NCT05165953
Title: Relationship Between Bronchial Asthma and COVID-19 Infection in Adults: Clinical and Laboratory Assessment
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, AMIRA HUSSEIN ALLAM, assistant professor of chest diseases and tuberculosis, Benha University
Other Study IDs: TEJB-D-21-00113
Record Dates: First submitted 2021-12-11; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Asthma; COVID-19
MeSH Terms: conditions — Asthma; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: COVID-19 positive with asthma: data were collected from medical records including: history of COVID -19 infection, presenting symptoms and clinical examination, hospitalization either ICU or ward. For asthma patients, their full data were collected regarding asthma control in last 3 months following GINA criteria for asthma control [8], Investigations included; CBC with differential count, WBC, lymphocytes, eosinophils, HGB and platelets, Inflammatory markers as d-dimer, LDH and ferritin level, electrolytes, BUN, serum creatinine, CXR, and old spirometry reports.
  Diagnosis of COVID 19 infection was made by a positive nasopharyngeal and throat swabs COVID 19 polymerase chain reaction (PCR).
  Interventions: Other: no intervention
- Group 2: COVID-19 positive with no asthma: data were collected from medical records including: history of COVID -19 infection, presenting symptoms and clinical examination, hospitalization either ICU or ward. Investigations included; CBC with differential count, WBC, lymphocytes, eosinophils, HGB and platelets, Inflammatory markers as d-dimer, LDH and ferritin level, electrolytes, BUN, serum creatinine, CXR, and old spirometry reports.
  Diagnosis of COVID 19 infection was made by a positive nasopharyngeal and throat swabs COVID 19 polymerase chain reaction (PCR).
  Interventions: Other: no intervention
- Group 3: COVID-19 negative with asthma: data were collected from medical records including: history of COVID -19 infection, presenting symptoms and clinical examination, hospitalization either ICU or ward. For asthma patients, their full data were collected regarding asthma control in last 3 months following GINA criteria for asthma control [8], Investigations included; CBC with differential count, WBC, lymphocytes, eosinophils, HGB and platelets, Inflammatory markers as d-dimer, LDH and ferritin level, electrolytes, BUN, serum creatinine, CXR, and old spirometry reports.
  Diagnosis of COVID 19 infection was made by a positive nasopharyngeal and throat swabs COVID 19 polymerase chain reaction (PCR).
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — there was no intervention in the study

SUMMARY:
Background: Asthma is still considered a major chronic respiratory disease that affects a large number in the world. The association between COVID-19 infection and asthma was studied in different ways focusing on hospital admitted patients. This study aimed to evaluate the relation between asthma and COVID-19 infection in adults attending outpatient pulmonary clinic over three successive months from clinical and laboratory point of view. Patients and methods: The current study collected 1309 patients attending the outpatient pulmonary clinic of a Saudi Arabian private Hospital over three successive months from 1st of December 2020 to the end of February 2021. Patients were divided into three groups; Group 1: COVID-19 infected with asthma (312), Group 2: COVID-19 infected with no asthma (286) and Group 3: COVID-19 non-infected with asthma (300).

DETAILED DESCRIPTION:
The current study aimed to evaluate the relation between asthma and COVID-19 infection in adults attending outpatient pulmonary clinic over three successive months from clinical and laboratory point of view.

Patients and methods:

The current study is a retrospective analytical study on 1309 patients attending pulmonary clinic in a Saudi Arabian private hospital over three successive month's starting from the 1st of December 2020 to the end of February 2021. Patients were classified according to previous history of asthma and /or infection with covid -19 in the previous 6 months. Patients were divided into two main groups according to history of COVID-19 infection; history of COVID-19 infection , no history of COVID-19 infection. Each group was divided into asthma and non-asthma groups. Patients who had no history of asthma and had no history of previous infection with COVID-19 were excluded from the study. So, the investigators get three groups: Group 1: COVID-19 positive with asthma, Group 2: COVID-19 positive with no asthma and Group 3: COVID-19 negative with asthma. The study was approved by local internal ethics committee and patient's acceptance to reveal their data was received prior to the study.

Methods: data were collected from medical records including: history of COVID -19 infection, presenting symptoms and clinical examination, hospitalization either ICU or ward. For asthma patients, their full data were collected regarding asthma control in last 3 months following GINA criteria for asthma control [8], Investigations included; CBC with differential count, WBC, lymphocytes, eosinophils, HGB and platelets, Inflammatory markers as d-dimer, LDH and ferritin level, electrolytes, BUN, serum creatinine, CXR, and old spirometry reports.

Diagnosis of COVID 19 infection was made by a positive nasopharyngeal and throat swabs COVID 19 polymerase chain reaction (PCR). The data were collected from patients' medical records including medical history, demographic information such as age, gender, symptoms of COVID-19, time of onset of symptoms, the physical examination at admission, during hospitalization, medications prescribed for COIVID-19 treatment, laboratory examinations, and imaging tests which were performed for all groups.

The data were analyzed using SPSS 22 (SPSS Inc., Chicago, IL, USA). The results were presented as percentile (absolute numbers); mean and standard deviation. Quantitative data were presented as median (interquartile range) (IQR, presented as first quartile - third quartile). Qualitative data were expressed as percentage (%) [9].

ELIGIBILITY:
Inclusion Criteria: patients with diagnosis of COVID19 infection in the past 6month and/or patient with diagnosis of asthma

Exclusion Criteria:

* patients with no history of COVID or asthma
* other diagnoses as cardiac or COPD or bronchiectasis, tuberculosis etc

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were classified according to previous history of asthma and /or infection with covid -19 in the previous 6 months. Patients were divided into two main groups according to history of COVID-19 infection; history of COVID-19 infection , no history of COVID-19 infection. Each group was divided into asthma and non-asthma groups. Patients who had no history of asthma and had no history of previous infection with COVID-19 were excluded from the study. So, we get three groups: Group 1: COVID-19 positive with asthma, Group 2: COVID-19 positive with no asthma and Group 3: COVID-19 negative with asthma.
Sampling Method: Non-Probability Sample
Enrollment: 1309 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
asthma control | 3 month
  study difference in asthma control between COVID and non COVID patients

SECONDARY OUTCOMES:
difference between groups | 3 month
  compare clinical and laboratory difference in parameters between the 3 groups

CONTACTS AND LOCATIONS:
Locations (1):
- RAFA medical centre, Riyāḑ, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
all collected data
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after acceptance by journal, for 1 year